CLINICAL TRIAL: NCT06252753
Title: An Observational Multi Center Study to Evaluate Real World Treatment Outcomes of Durvalumab Based Regimens in Hepatobiliary Cancers
Brief Title: Observational Study Protocol: LIVER-R
Acronym: LIVER-R
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Other Study IDs: D419CR00035
Record Dates: First submitted 2023-12-21; First posted 2024-02-12 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Hepatobiliary Cancers
Keywords: Hepatobiliary cancer; Unresectable hepatocellular carcinoma (uHCC); Advanced biliary tract cancer (aBTC); Durvalumab; Observatory; Real-world
MeSH Terms: interventions — durvalumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- unresectable hepatocellular carcinoma (uHCC): unresectable hepatocellular carcinoma (uHCC)
  Interventions: Other: Durvalumab-based combination therapies in observational study setting
- advanced biliary tract cancer (aBTC): advanced biliary tract cancer (aBTC)
  Interventions: Other: Durvalumab-based combination therapies in observational study setting

INTERVENTIONS:
Other: Durvalumab-based combination therapies in observational study setting — Data on patients who initiated durvalumab-based regimens, including STRIDE (Single Tremelimumab Regular Interval Durvalumab), will be collected).
  Other Names: Imfinzi
  Groups: unresectable hepatocellular carcinoma (uHCC)
Other: Durvalumab-based combination therapies in observational study setting — Data on patients who initiated durvalumab-based regimens, including durvalumab + chemotherapy combinations (e.g., Durvalumab + GemCis etc.) will be collected.
  Other Names: Imfinzi
  Groups: advanced biliary tract cancer (aBTC)

SUMMARY:
Given the number of anticipated durvalumab-based treatment launches in the hepatobiliary cancer space over the next 3 years, there is a need to capture contemporary real-world data across these indications. LIVER-R is a multicountry, multicenter, observational study of patients with a confirmed diagnosis of hepatobiliary cancer treated with a durvalumab-based regimen as part of routine clinical practice or early access program (EAP). The study design will include primary and secondary data collection. The primary objective of this study is to evaluate the effectiveness of durvalumab-based regimens in real-world settings as measured by real-world overall survival. Other endpoints include demographics, clinical characteristics, clinically significant events of interest, treatment patterns, concomitant medications, and other real-world clinical endpoints (such as duration of treatment, progression-free survival, time to treatment progression, time to next treatment, recurrence-free survival, and time to treatment recurrence).

DETAILED DESCRIPTION:
LIVER-R is a real-world, multi-country, multi-centre study aiming to enroll approximately 2500 pts with unresectable hepatocellular carcinoma (uHCC; n=1135) or advanced biliary tract cancers (aBTCs; n=1355) across 22 countries from North and South America, Europe, the Middle East and the Asia-Pacific region. The study design will include primary and secondary data collection. Primary data will be collected in real-time during the patient's routine visit. Secondary data will be collected from the patient's medical record at enrollment and at prespecified study time points (6-month intervals). The study population includes adult patients whose physician has previously made the decision to treat them with a durvalumab-based regimen for hepatobiliary cancer as part of routine clinical practice or patients receiving treatment through EAP. The study will include a baseline period of up to 5 years before the index date (initiation of a Durvalumab-based regimen) and a follow-up period to the earliest of death, loss to follow-up, withdrawal, or end of study for a maximum follow-up of 2 years for patients with aBTCs or 3 years for patients with uHCC. This is a descriptive, noncomparative study. No formal hypotheses are to be tested. All descriptive analyses will be conducted separately for each primary hepatobiliary cancer indication. Kaplan Meier estimates will be produced for time-to-event outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and a lawful adult in the country at the index date
2. Confirmed presence of malignancy of primary hepatobiliary cancer (i.e., uHCC or aBTC) by the treating physician
3. Type of hepatobiliary cancer indication is approved to be treated (i.e., positive phase 3 clinical trial read out for HIMALAYA or TOPAZ 1) with a durvalumab based regimen in the respective country or was administered as part of an EAP
4. Informed consent was obtained as per country level regulations on or after the index date

Exclusion Criteria:

1. Currently/was participating or plans to participate in any clinical trial for investigational treatment for hepatobiliary cancers on or after the diagnosis date until the index date
2. Received other systemic therapies for hepatobiliary cancer indication on or after diagnosis date through the index date (e.g., uHCC or aBTC patient who received a systemic treatment for unresectable HCC or advanced BTC, respectively, prior to initiating durvalumab based regimen)
3. Received a liver transplant during the baseline period

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients treated with a durvalumab based regimen for hepatobiliary cancer as part of routine clinical practice. The decision to treat patients with a durvalumab based regimen should be independent from the decision to enroll patients in the study. Depending on the country, it is anticipated that 15 to 400 patients may be enrolled in each participating country.
Sampling Method: Non-Probability Sample
Enrollment: 4490 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Real-world overall survival (rwOS) | rwOS will be assessed as OS rates at 6, 12, 24 months (both aBTC and uHCC), and 36 months (uHCC), median OS for a maximum follow-up of 2 and 3 years for aBTC and uHCC, respectively.
  rwOS will be calculated as the time from the index date to date of death, by any cause.

SECONDARY OUTCOMES:
Real-world duration of treatment (rwDOT) | rwDOT will be assessed as median DOT for a maximum follow-up of 2 years (aBTC) or 3 years (uHCC).
  rwDOT will be calculated for each systemic treatment as the time from the index date to date of discontinuation for any reason.
Real-world progression free survival (rwPFS) | rwPFS will be assessed as PFS rates at 6, 12, 24 months (both aBTC and uHCC), and 36 months (uHCC), median PFS for a maximum follow-up of 2 and 3 years for aBTC and uHCC, respectively.
  rwPFS will be calculated as the time from the index date to the date of documented disease progression as determined by the physician's assessment or death, whichever is earlier.
Real-world time to progression (rwTTP) | rwTTP will be assessed as median TTP for a maximum follow-up of 2 years (aBTC) or 3 years (uHCC).
  rwTTP will be calculated as the time from the index date to the date of documented disease progression as determined by the physician's assessment.
Real-world time to next treatment (rwTTNT) | rwTTNT will be assessed as median TTNT for a maximum follow-up of 2 years (aBTC) or 3 years (uHCC).
  rwTTNT will be calculated as the time from the index date to the date of initiation of the next treatment.
Real-world recurrence free survival (rwRFS) | rwRFS will be assessed as RFS rates at 6, 12, 24 months (both aBTC and uHCC), and 36 months (uHCC), median RFS for a maximum follow-up of 2 and 3 years for aBTC and uHCC, respectively.
  rwRFS will be defined as the time from the index date to the date of documented disease recurrence as determined by the physician's assessment or death, whichever is earlier. The analysis will be performed in patients who underwent curative therapy (resection or ablation).
Real-world time to recurrence (rwTTR) | rwTTR will be assessed as median TTR for a maximum follow-up of 2 years (aBTC) or 3 years (uHCC).
  rwTTR will be defined as the time from the index date to the date of documented disease recurrence as determined by the physician's assessment. The analysis will be performed in patients who underwent curative therapy (resection or ablation).
Patient demographic and clinical characteristics | Patient demographic and clinical characteristics will be captured up to 5 years prior to the index date.
  Descriptive statistics will be used to describe demographic and clinical characteristics for the enrolled patients.
Percentage of patients receiving each treatment regimen | Treatment patterns will be captured from the index date until the earliest of death, loss to follow-up, withdrawal, or end of study for a maximum follow-up of 2 years for patients with aBTCs or 3 years for patients with uHCC.
  Treatment patterns will be calculated from the index date until death, loss to follow-up, withdrawal from the study, or end of the study, whichever is earliest.
Clinically significant events (CSEs) of interest leading to a medical intervention | CSEs will be captured from the index date through 90 days after the last administration of durvalumab-based regimen or death, whichever occurs first.
  CSEs of interest leading to medical intervention including durvalumab based treatment interruption, discontinuation, hospitalization, or which require interventions of concomitant use of corticosteroids, immunosuppressants and/or endocrine therapies will be captured for the enrolled patients.

CONTACTS AND LOCATIONS:
Locations (126):
- United States (21):
  - Research Site, Birmingham, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Coronado, California
  - Research Site, Los Angeles, California
  - Research Site, Walnut Creek, California
  - Research Site, Clermont, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Tampa, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Evergreen Park, Illinois
  - Research Site, Hinsdale, Illinois
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Osage Beach, Missouri
  - Research Site, White Plains, New York
  - Research Site, Canton, Ohio
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Dallas, Texas
  - Research Site, Temple, Texas
  - Research Site, Spokane, Washington
- Australia (4):
  - Research Site, Garran, Australian Capital Territory
  - Research Site, Heidelberg, Victoria
  - Research Site, Melbourne, Victoria
  - Research Site, Murdoch, Western Australia
- Austria (3):
  - Research Site, Sankt Pölten, Lower Austria
  - Research Site, Linz, Upper Austria
  - Research Site, Vienna, Vienna
- Belgium (6):
  - Research Site, Brussels, Anderlecht
  - Research Site, Bonheiden, Antwerp
  - Research Site, Edegem, Antwerp
  - Research Site, Leuven, Brabant
  - Research Site, Liège, Wallonia
  - Research Site, Stene, West Flanders
- Brazil (5):
  - Research Site, Curitiba, Paraná
  - Research Site, Recife - PE, Recife - PE
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, Morumbi, São Paulo
  - Research Site, São Paulo
- Research Site, Halifax, Nova Scotia, Canada
- France (9):
  - Research Site, Strasbourg, Alsace
  - Research Site, Grenoble, Auvergne-Rhône-Alpes
  - Research Site, St-Malo, Brittany Region
  - Research Site, Mulhouse, Grand Est
  - Research Site, Boulogne-sur-Mer, Hauts-de-France
  - Research Site, Poitiers, Nouvelle-Aquitaine
  - Research Site, Avignon, Provence-Alpes-Côte d'Azur Region
  - Research Site, Marseille, Provence-Alpes-Côte d'Azur Region
  - Research Site, Paris, Île-de-France Region
- Germany (26):
  - Research Site, Heidenheim, Baden W Rttemberg
  - Research Site, Konstanz, Baden-Wurttemberg
  - Research Site, Mannheim, Baden-Wurttemberg
  - Research Site, Schorndorf, Baden-Wurttemberg
  - Research Site, Stuttgart, Baden-Wurttemberg
  - Research Site, Augsburg, Bavaria
  - Research Site, Munich, Bavaria
  - Research Site, Bremenhaven, City state Bremen
  - Research Site, Kassel, Hesse
  - Research Site, Marburg, Hesse
  - Research Site, Wiesbaden, Hesse Land
  - Research Site, Göttingen, Lower Saxony
  - Research Site, Hanover, Lower Saxony
  - Research Site, Aachen, North Rhine-Westphalia
  - Research Site, Bochum, North Rhine-Westphalia
  - Research Site, Dortmund, North Rhine-Westphalia
  - Research Site, Moers, North Rhine-Westphalia
  - Research Site, Stolberg, North Rhine-Westphalia
  - Research Site, Koblenz, Rhineland-Palatinate
  - Research Site, Dresden, Saxony
  - Research Site, Leipzig, Saxony
  - Research Site, Halle, Saxony-Anhalt
  - Research Site, Magdeburg, Saxony-Anhalt
  - Research Site, Neumünster, Schleswig-Holstein
  - Research Site, Berlin
  - Research Site, Hamburg
- Greece (4):
  - Research Site, Chaïdári, Athens
  - Research Site, Athens, Attica
  - Research Site, Thessaloniki, Central Macedonia
  - Research Site, Larissa, Thessaly
- Israel (4):
  - Research Site, Nahariya, Northern Didstrict
  - Research Site, Ramat Gan, Tel Aviv
  - Research Site, Jerusalem
  - Research Site, Tel Aviv
- Italy (8):
  - Research Site, Naples, Campania
  - Research Site, Rome, Lazio
  - Research Site, Brescia, Lombardy
  - Research Site, Milan, Lombardy
  - Research Site, Rozzano, Lombardy
  - Research Site, Turin, Piedmont
  - Research Site, Monserrato, Sardinia
  - Research Site, Pisa, Tuscany
- Japan (8):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Kashiwa-shi, Chiba
  - Research Site, Kurume, Fukuoka
  - Research Site, Kanazawa, Ishikawa-ken
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kyoto, Kyoto
  - Research Site, Sendai, Miyagi
  - Research Site, Ōsaka-sayama, Osaka
- Research Site, Lisbon, Portugal
- Research Site, San Juan, Rio Piedras, Puerto Rico
- Romania (3):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Iași
- Saudi Arabia (2):
  - Research Site, Riyadh, Ar Riyadh
  - Research Site, Jeddah, Mecca Region
- Research Site, Singapore, Singapore
- Spain (14):
  - Research Site, Santiago de Compostela, A Coruna
  - Research Site, Zaragoza, Aragon
  - Research Site, Santander, Cantabria
  - Research Site, Burgos, Castille and León
  - Research Site, Poniente Sur, Cordoba
  - Research Site, Ourense, Galicia
  - Research Site, El Palmar, Murcia
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Oviedo
  - Research Site, Pamplona
  - Research Site, Santa Cruz de Tenerife
  - Research Site, Seville
  - Research Site, Valencia
- Research Site, Zurich, Switzerland
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Taipei
  - Research Site, Taoyuan
- Research Site, Mohammed Bin Zayed City, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
Plan to share only the redacted CSR synopsis
Supporting Information: CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Derived] Ikeda M, Worns MA, Akce M, Hsu C, Tebbutt NC, Casadei-Gardini A, Sah J, Farid-Kapadia M, Stirnadel-Farrant HA, Paskow MJ, Baur B, Melillo G, Schmidt J, Daktera A, Knox JJ. LIVER-R study protocol: a global real-world study of durvalumab-based regimens in patients with hepatobiliary cancers. Future Oncol. 2025 Dec;21(29):3739-3748. doi: 10.1080/14796694.2025.2589057. Epub 2025 Nov 24. PMID 41277677